CLINICAL TRIAL: NCT04376073
Title: An Open-label, Single Arm, Phase II Trial of Niraparib in Combination With Anlotinib in Patients With Platinum-resistant Recurrent Ovarian Cancer, Fallopian Tube Cancer, and Primary Peritoneal Cancer (Ovarian Cancer)
Brief Title: Anlotinib and Niraparib Dual Therapy Evaluation in Platinum-resistant Recurrent Ovarian Cancer
Acronym: ANNIE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jihong Liu (Other)
Responsible Party: Sponsor-Investigator, Jihong Liu, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-FXY-357
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Platinum-resistant Ovarian Cancer
MeSH Terms: interventions — niraparib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Niraparib 300mg(Body Weigh ≥77 kg)/200mg (Body Weigh <77 kg) po QD day1~21, Anlotinib 12mg po QD day1~14.
  Starting dose of anlotinib changed to 10mg from 2020-11-13.
  Interventions: Drug: Niraparib; Drug: Anlotinib

INTERVENTIONS:
Drug: Niraparib — Niraparib 300mg(Body Weigh ≥77 kg)/200mg (Body Weigh <77 kg) po QD day1~21, Anlotinib 12mg po QD day1~14
Drug: Anlotinib — Anlotinib 12mg po QD day1~14. Starting dose of anlotinib changed to 10mg from 2020-11-13.

SUMMARY:
At present, the standard treatment for platinum-resistant ovarian cancer patients is platinum-free chemotherapy, with poor efficacy and tolerance. The combination of anti-angiogenic drugs and PARPi can play a synergistic anti-tumor role and achieve good efficacy in platinum-sensitive recurrent ovarian cancer. This study intends to explore the safety and effectiveness of anlotinib and niraparib dual therapy in patients with platinum-resistant recurrent ovarian cancer, fallopian tube cancer, and primary peritoneal cancer (ovarian cancer).

DETAILED DESCRIPTION:
The present study is an open, single-center, prospective, single-arm phase II study to investigate the efficacy and safety of nilapalil combined with anrotidine in the treatment of platinum-resistant recurrent ovarian cancer. In this study, 40 histopathologically diagnosed patients with high-grade serous ovarian, fallopian tube and primary peritoneal cancer were treated with neelapalil plus anrotinib in patients who underwent first-line chemotherapy or above and had a recurrence of platinum-resistant chemotherapy (the time of tumor progression of the last platinum-containing chemotherapy < 6 months). The study will be divided into two phases. The first phase will include six patients on a 21-day cycle (nierapalil 200mg QD*21; Anrotidine 12mg qd d1-14, d15-21 suspension), all subsequent patients were enrolled if no more than dose-restricted toxic event occurred within a cycle, and the combination treatment was continued until the disease progressed or the toxicity was intolerable.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects understand the trial process, sign informed consent, agree to participate in the study, and have the ability to follow the protocol; 2. 18 ~ 70 years old (inclusive), female; 3. Histologically diagnosed ovarian, fallopian tube, or primary peritoneal cancer; 4. Subjects were initially treated with platinum, and the disease recurrence occurred within 6 months after the end of the previous platinum-containing chemotherapy, that is, platinum resistance relapsed; 5. Life expectancy > 16 weeks; 6. Patient's ECOG physical status score is 0-1; 7. Subject agrees to take blood samples for gBRCA mutations; 8. Can provide formalin-fixed, paraffin-embedded tumor tissue samples for sBRCA and homologous recombination repair-related genes detection (optional); 9. Good organ function, including:
* Neutrophil count >= 1500 / μL;
* Platelets >= 100,000 / μL;
* Hemoglobin >= 9g / dL;
* Serum creatinine <= 1.5 times the upper limit of normal value, or creatinine clearance >= 60mL / min (calculated according to Cockcroft-Gault formula);
* Total bilirubin <= 1.5 times the upper limit of normal value or direct bilirubin <= 1.0 times the upper limit of normal value;
* AST and ALT <= 2.5 times the upper limit of normal value. When liver metastases are present, it must be <= 5 times the upper limit of normal value.

  10. The toxic side effects of any previous chemotherapy have recovered to <= CTCAE level 1 or baseline levels, except for sensory neuropathy or hair loss with stable symptoms <= CTCAE level 2.

Exclusion Criteria:

1. People who are known to be allergic to Niraparib or Anlotinib (or active or inactive ingredients of drugs with similar chemical structure);
2. Symptomatic, uncontrolled brain or pia mater metastases;
3. Underwent major surgery within 3 weeks before the study began or has not recovered after surgery;
4. Received palliative radiotherapy of > 20% bone marrow 1 week before enrollment;
5. Have invasive cancer other than ovarian cancer (except fully treated basal or squamous cell skin cancer) within 2 years before enrollment;
6. Patients with central lung squamous cell carcinoma or at risk for large hemoptysis;
7. Previous or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
8. Severe or uncontrolled diseases, including but not limited to: uncontrollable nausea and vomiting, inability to swallow or gastrointestinal diseases that may interfere with drug absorption and metabolism; active viral infections; mental illnesses that affect patients' signed informed consent History of bleeding tendency and thrombosis; history of severe cardiovascular disease;
9. Laboratory abnormalities: hyponatremia; hypokalemia; uncontrollable nail function abnormalities;
10. Receive platelet or red blood cell transfusions within 4 weeks;
11. Patients who are pregnant or nursing, or who plan to become pregnant during study treatment;
12. Have previously received any PARP inhibitor treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | at 6 months
  The primary objective of this study is to determine the preliminary efficacy of administration of niraparib in combination with anlotinib in the treatment of platinum-resistant recurrent ovarian cancer, as measured by the objective response rate (ORR), which is a combination of CR (the target lesion completely disappeared over 4 weeks) and PR (Target lesions were reduced by more than 30% for more than 4 weeks).

SECONDARY OUTCOMES:
The frequency and severity of adverse events | Baseline through 1 year
  The frequency and severity of adverse events and toxicity based upon NCI CTCAE version 5.0 during subjects receiving the study treatment.
Progression-free survival | at 6 months
  Progression-free survival is defined as the time from enrollment to first documentation of tumor progression, or to death due to any cause in the absence of previous documentation of objective tumor progression.
Objective tumor response | at 6 months
  The total proportion of subjects who have an objective tumor reponse (CR + PR) using the RECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within six months after the trial complete
URL: http://www.medresman.org.cn

REFERENCES:
- [Derived] Deng T, Yan L, Li J, Liu G, Yin A, Feng Y, Zheng M, Zhang C, Huang H, Huang Q, Lin A, Jiang J, Kong B, Liu J. Adverse Event Management in Patients with Platinum-Resistant Ovarian Cancer Treated with Niraparib and Anlotinib: Updates from the Phase II, Multi-Center ANNIE Study. Ther Clin Risk Manag. 2025 Jul 21;21:1135-1147. doi: 10.2147/TCRM.S526755. eCollection 2025. PMID 40718116
- [Derived] Liu G, Feng Y, Li J, Deng T, Yin A, Yan L, Zheng M, Xiong Y, Li J, Huang Y, Zhang C, Huang H, Wan T, Huang Q, Lin A, Jiang J, Kong B, Liu J. A novel combination of niraparib and anlotinib in platinum-resistant ovarian cancer: Efficacy and safety results from the phase II, multi-center ANNIE study. EClinicalMedicine. 2022 Nov 30;54:101767. doi: 10.1016/j.eclinm.2022.101767. eCollection 2022 Dec. PMID 36583171